CLINICAL TRIAL: NCT05854914
Title: Benefit of Hypnosis on Smartphone for Acute Post-operative Pain
Brief Title: Benefit of Hypnosis on Smartphone for Acute Post-operative Pain (HYPNO-APP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-AOIP-05
Record Dates: First submitted 2023-04-27; First posted 2023-05-11 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Appendicitis With Peritonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypnosis video to control postoperative pain. (Experimental)
  Interventions: Procedure: Use of hypnosis videos

INTERVENTIONS:
Procedure: Use of hypnosis videos — Hypnosis on smartphone will be used to manage pain for emergent coelioscopy surgery of patients with acute and complicated appendicitis, with generalized peritonitis

SUMMARY:
Appendicitis is a common pathology and the one of the most common surgical procedures performed in France. Young subjects are the most frequent patients with appendicitis. Appendicular peritonitis increases post-operative pain, morbidity, and the average length of hospital stay compared to uncomplicated appendicitis.

Pain alters perioeprative rehabilitation of patients. Surgery, performed urgently, generates more anxiety and pain than scheduled surgery. But, intensity of chronic postoperative pain is in correlation to intensity of acute postoperative pain. In addition, admission of emergency cases is more axiety-inducing, due to wait times, packed emergency room, worklaod of medical staff.

Sex and age also modify perception of postoperative pain. Adults under 50 feel more pain than older patients for similar procedures.

Medication for pain is required in perioperative period et is administered according protocol of each medical center ; these protocols include analgesics, opioids or not, benzodiazepine... However, opioids analgesic (example: morphine) can induce side effect, such as confusional syndrome, cardio-pulmonary manifestations, ileus, nausea and vomiting...

Non-pharmacological approaches have been also proposed to reduce anxiety and pain. Hypnosis is frequently used but not always adapted to the emergency: need for qualified and available staff, environment not conducive to hypnotic induction...

Hypnosis is a modified state of consciousness ; it is neither a state of vigilance nor a state of sleep. Several types of hypnosis can be distinguished according to the medical application, such as hypnoanalgesia or hypnosedation.

Using hypnosedation during surgical or invasive procedure can reduce the use of painkillers and sedatives. Interest of hypnosis has been observed for extraction of wisdow teeth, delivery...

Young patients are very comfortable with the use of their smartphone which is often the first object recovered when they return from the operating room. Many hypnosis videos are available free of charge on Internet, and some of which are produced by specialized practitioners and university teachers.

A recent study has shown that among young people, addiction to smartphone is a predisposition to hypnosis.

However, the use of hypnosis videos on smartphone has never been studied for the control of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Complicated acute appendicitis with generalized appendicitis, coelioscopy emergency surgery
* Signature of the written informed consent form by the patient
* Affiliation to a French health insurance scheme or equivalent
* Patient inderstands French and has a smartphone with internet access

Non inclusion Criteria:

* Uncomplicated or complicated appendicitis of abscesses, presence of an intraperitoneal abscess, a plastron, uncomplicated appendicitis of generalized peritonitis
* Patient with a neurological, visual or auditory condition where videos cannot be viewed
* Presence of active cancer, a malignant hemopathy, drug addiction, coagulopathy, immunosuppressive treatment
* Non-acute or interval appendectomy, i.e. after antibiotic treatment of a complicated appendicitis of the plastron or drainage of an appendicular abscess;
* Vulnerable people: adult under guardianship, curator ship or deprived of freedom.
* Medication or pathology affecting ability to discern: Severe psychotic disorders
* Patient refusing to monitor anxiety and pain via smartphone
* Patient already medically monitored for anxiety, depressive or chronic pain syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To study the effect of hypnosis on smartphone on postoperative pain in patients operated in emergency by coelioscopy of acute and complicated appendicitis with peritonitis. | During the first postoperative week
  Efficacy of hypnosis on smartphone will be defined by the evolution of pain. Pain will be measured with a visual and analogic scale, before and after each hypnosis session. The scame ranges from 0 (no pain) to 10 (maximum thinkable pain).

SECONDARY OUTCOMES:
To study the effect of hypnosis on smartphone on the use of analgesics during hospitalization. | 30 days post surgery
  A standardized analgesic protocol is implemented in order to each patient receives painkillers in the same way after inclusion. The amount of morphine received during hospitalization will be expressed as morphine equivalent.
To study the effect of hypnosis on smartphone on the average length of hospital stay after the beginning of hypnosis sessions | 30 days post surgery
  The length of hospitalization is the cumulative length of the entire hospital stay(s) in days until the 30th postoperative day (rehospitalizations included). The length of stay in a non-hospital health structure, such as a convalescent center, will not be included.
To study the effect of hypnosis on smartphone on the anxiety before and after hypnosis sessions | At inclusion and 2 days after inclusion
  Anxiety will be measured using the Anxiety-State scale from Spielberger. It assesses the feelings of apprehension, tension, nervousness and worry that the subject feels at the time of the anxiety or the competitive situation. This questionnaire is an indicator of transient changes in anxiety caused by adverse or therapeutic situations. For each question, answers are ranged from 1 to 4. If the total score exceeds 51 for men, 61 for women, the patient is considered anxious.
To study the effect of hypnosis on smartphone on morbidity at postoperative day 30. | 30 days post surgery
  Morbidity will be classified according to the Clavien-Dindo classification. This classification was originally published in 2004 in the Annals of Surgery for elective general surgery. Later, it has been objectively validated for all surgical specialties. This classification ranks complications from 0 (no complication) to 5 (death).

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No